CLINICAL TRIAL: NCT00004103
Title: A Phase II Study of Systemic Therapy With CPT-11 (Camptosar HCl) and Cisplatin in Patients With Advanced Gastric Cancer to be Followed by Surgical Resection and Postoperative Intraperitoneal Chemotherapy
Brief Title: Combination Chemotherapy Followed by Surgery in Treating Patients With Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067322; P30CA016087 (NIH); NYU-9822; P-UPJOHN-647597196; NCI-G99-1594
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Gastric Cancer
Keywords: stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Floxuridine; Irinotecan; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: floxuridine
Drug: irinotecan hydrochloride
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and combining chemotherapy with surgery may kill more tumor cells.

PURPOSE: This phase II trial is studying how well irinotecan and cisplatin followed by surgery, floxuridine, and cisplatin work in treating patients with stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete and partial response rates and time to treatment failure in patients with advanced gastric cancer treated with neoadjuvant irinotecan and cisplatin followed by surgery then intraperitoneal floxuridine and cisplatin.
* Determine the rate of potentially curative surgery in patients receiving this regimen.
* Determine the toxicity and tolerance of this regimen in these patients.

OUTLINE: Patients receive cisplatin IV and irinotecan IV once a week for 4 weeks. This course is repeated 2 weeks later.

Patients who achieve complete or partial remission or stable disease undergo resection 4 weeks after the last chemotherapy dose.

Patients with no residual macroscopic disease begin adjuvant intraperitoneal (IP) chemotherapy 1 week after surgery. Chemotherapy consists of floxuridine IP over 30 minutes on days 1-3 and days 22-24 and cisplatin IP on days 3 and 24.

PROJECTED ACCRUAL: A total of 18-33 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven, previously untreated gastric cancer

  * Stage IB, II, III, or IV (T3-4, N0 OR any T, N1-2, M0)
  * No metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin less than 2 mg/dL
* SGOT/SGPT no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 3 times ULN
* PT, aPTT, and TT normal
* No Gilbert's disease

Renal:

* BUN no greater than 30 mg/dL
* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No myocardial infarction within the past 3 months
* No congestive heart failure requiring therapy

Other:

* No other invasive malignancy in the past 5 years except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* No active or uncontrolled infection
* HIV negative
* No other severe concurrent disease
* No psychiatric disorders that would preclude compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for gastric cancer

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for gastric cancer

Surgery:

* No prior surgery for gastric cancer
* No emergent need for surgery for gastrointestinal obstruction, perforation, or hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-07; Primary Completion 2007-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Newman, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU Cancer Institute at New York University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Newman E, Potmesil M, Ryan T, Marcus S, Hiotis S, Yee H, Norwood B, Wendell M, Muggia F, Hochster H. Neoadjuvant chemotherapy, surgery, and adjuvant intraperitoneal chemotherapy in patients with locally advanced gastric or gastroesophageal junction carcinoma: a phase II study. Semin Oncol. 2005 Dec;32(6 Suppl 9):S97-100. doi: 10.1053/j.seminoncol.2005.06.002. PMID 16399443